CLINICAL TRIAL: NCT04542525
Title: Clinical Investigation of AcrySof IQ PanOptix Toric Intraocular Lens Model TFNT20
Brief Title: Clinical Investigation of an AcrySof IQ PanOptix Toric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILX140-C001
Record Dates: First submitted 2020-09-03; First posted 2020-09-09 (Actual); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-07

CONDITIONS: Aphakia; Corneal Astigmatism
Keywords: Cataract; Intraocular lens; Astigmatism; Toric
MeSH Terms: conditions — Aphakia; Astigmatism; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- PanOptix Toric Trifocal IOL (Experimental): ACRYSOF IQ PanOptix Toric Trifocal IOL Model TFNT20 implanted in the capsular bag in the posterior chamber following cataract surgery. At least one eye will be implanted.
  Interventions: Device: ACRYSOF IQ PanOptix Toric Trifocal IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: ACRYSOF IQ PanOptix Toric Trifocal IOL — Single-piece, ultraviolet and blue-light filtering, foldable, multifocal toric IOL intended to provide vision to aphakic subjects at near, intermediate, and distance and to correct pre-existing corneal astigmatism
  Other Names: PanOptix Toric Trifocal IOL; Model TFNT20
Procedure: Cataract surgery — Cataract extraction by phacoemulsification, followed by implantation of the IOL per investigator's standard of care and instructions for use

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the TFNT20 low cylinder power intraocular lens when implanted in the eye to replace the natural lens following cataract removal.

DETAILED DESCRIPTION:
Subjects will attend a total of 5 to 9 visits, depending on whether one eye or both eyes are implanted. The second eye surgery, if applicable, will occur 1 to 30 days after the first eye surgery. Total individual duration of participation will be up to 4 months, including an up to 2-month preoperative period.

This study will be conducted in Japan.

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible to be implanted with AcrySof IQ PanOptix Toric Intraocular Lens Model TFNT20 in at least one eye.
* Potential postoperative Best Corrected Distance Visual Acuity (BCDVA) of 0.5 decimal or better.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Irregular corneal astigmatism.
* History of anterior segment, posterior segment, or optic nerve pathology.
* History of previous intraocular or corneal (refractive or trauma related) surgery.
* Any other planned ocular surgical procedures including but not limited to limbal relaxing incision (LRI)/Astigmatic Keratotomy and laser assisted in situ keratomileusis (LASIK).
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Japan Limited
Locations (1):
- Alcon Investigative Site, Chiyoda-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 investigative site located in Japan.
Pre-assignment Details: This reporting group includes all enrolled participants.
Units Other Than Participants: eyes
Groups:
- PanOptix Toric Trifocal IOL: ACRYSOF IQ PanOptix Toric Trifocal IOL Model TFNT20 implanted in the capsular bag in the posterior chamber following cataract surgery
Period: Overall Study
Arm/Group | PanOptix Toric Trifocal IOL
Started | 32; 41 eyes
Attempted Implantation | 32; 41 eyes
Successful Implantation | 32; 41 eyes
Completed | 32; 41 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: All Implanted Analysis Set: All eyes with successful test article implantation
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.4)
Age, Customized [Number; unit: participants]
  Less than 60 years | 8
  60-69 years | 10
  70-79 years | 13
  80 years and older | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 32
Region of Enrollment [Number; unit: participants]
  Japan | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With ≤ 0.25 Diopter (D) Absolute Refractive Cylinder at Visit 3/3A (Day 30-60)
Description: A manifest refraction (manual vision test) was conducted using charts. Refractive cylinder is the amount of power in diopters that is needed to correct any remaining astigmatism.
Time Frame: Day 30-60 postoperative
Population: All Implanted Analysis Set
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 32
Number analyzed (eyes) | 41
percentage of eyes | 90.2
Statistical Analysis 1: Comparison: PanOptix Toric Trifocal IOL; Test type: Superiority; p < 0.0001, Exact Test of Binomial Proportion; P-value is provided from exact test of binomial proportion (one-sided alpha = 2.5%) comparing PanOptix Toric Trifocal IOL Model TFNT20 with historical threshold 29.2 % (rate calculated for a non-toric IOL in Japanese study patients that would qualify for a T2 lens using the same toric calculator)

2. Secondary Outcome: Percentage of Eyes With ≤ 0.5 Diopter (D) Absolute Refractive Cylinder at Visit 3/3A (Day 30-60)
Description: A manifest refraction (manual vision test) was conducted using charts. Refractive cylinder is the amount of power in diopters that is needed to correct any remaining astigmatism. No confirmatory statistical hypothesis testing was pre-specified in the protocol.
Time Frame: Day 30-60 postoperative
Population: All Implanted Analysis Set
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 32
Number analyzed (eyes) | 41
percentage of eyes | 100

3. Secondary Outcome: Average Absolute Manifest Refractive Cylinder at Visit 3/3A (Day 30-60)
Description: as for outcome 2
Time Frame: Day 30-60 postoperative
Population: All Implanted Analysis Set
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 32
Number analyzed (eyes) | 41
diopter | 0.055 (0.153)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected pre-treatment (Day -60 to 0) up to Day 30-60 post-treatment/study exit. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: This analysis population includes all subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye). "At Risk" population of pre-treatment and systemic AEs is reported in units of subjects; ocular AE population is reported in units of eyes.
Groups:
- Pretreatment: Events reported in this group occurred prior to attempted implantation with the test article
- TFNT20 Ocular / First Eye; TFNT20 Ocular / Second Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the study eye
- TFNT20 Nonocular / Systemic: Events reported in this group occurred after attempted implantation with the test article
Arm/Group | Pretreatment | TFNT20 Ocular / First Eye | TFNT20 Ocular / Second Eye | TFNT20 Nonocular / Systemic
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/9 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/9 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 5/32 | 1/9 | 0/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=32) | TFNT20 Ocular / First Eye (N=32) | TFNT20 Ocular / Second Eye (N=9) | TFNT20 Nonocular / Systemic (N=32)
Intraocular pressure increased (Investigations) | 0 | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT04542525/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT04542525/SAP_001.pdf